CLINICAL TRIAL: NCT02805348
Title: Long-Term Specified Drug Use-Results Survey in Patients With Pre-dialysis Chronic Kidney Disease
Brief Title: Post-marketing Surveillance of Bixalomer in Patients With Pre-dialysis Chronic Kidney Disease
Status: Completed | Type: Observational
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: 1585-MA-3052
Record Dates: First submitted 2016-06-16; First posted 2016-06-20 (Estimated); Last update posted 2024-10-16 (Actual); Status verified 2019-04

CONDITIONS: Chronic Kidney Disease
Keywords: Kiklin; Bixalomer; Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — bixalomer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chronic kidney disease: Patients with pre-dialysis chronic kidney disease complicated by hyperphosphatemia who used bixalomer for the first time.
  Interventions: Drug: Bixalomer

INTERVENTIONS:
Drug: Bixalomer — Oral
  Other Names: ASP1585; AMG223; Kiklin; ILY101

SUMMARY:
The objective of this study is to assess the long-term safety and efficacy of bixalomer under post-marketed setting.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pre-dialysis chronic kidney disease complicated by hyperphosphatemia who used bixalomer for the first time

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with pre-dialysis chronic kidney disease complicated by hyperphosphatemia who used bixalomer for the first time
Sampling Method: Non-Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the serum concentrations of phosphate | Baseline and up to Month 12
Change from baseline in the corrected serum concentrations of calcium | Baseline and up to Month 12
Change from baseline in the serum concentrations of intact parathyroid hormone | Baseline and up to Month 12
Safety assessed by incidence of adverse events | Up to Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Director — Astellas Pharma Inc
Locations (14):
- Japan (14):
  - Site JP00006, Aichi
  - Site JP00010, Ehime
  - Site JP00012, Fukuoka
  - Site JP00004, Gifu
  - Site JP00001, Ibaraki
  - Site JP00009, Kagawa
  - Site JP00003, Kanagawa
  - Site JP00011, Kochi
  - Site JP00014, Kumamoto
  - Site JP00013, Nagasaki
  - Site JP00007, Osaka
  - Site JP00005, Shizuoka
  - Site JP00002, Tochigi
  - Site JP00008, Wakayama

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.